CLINICAL TRIAL: NCT00412087
Title: Vitamin D Status of Pregnant Women and Their Children in Eau Claire, South Carolina: A Prevalence and Supplementation Model for Community Health Care Centers in the U.S.
Brief Title: Vitamin D Status of Pregnant Women and Their Children in Eau Claire, South Carolina
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Carol Wagner, Professor of Pediatrics, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HR-16476
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Vitamin D Deficiency; Pregnancy
Keywords: vitamin D; cholecalciferol; pregnant women
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cholecalciferol 2000 IU (Experimental): Women at 12-16 weeks' gestation are enrolled into the study to receive 2000 IU/day vitamin D3 for one month. After the run-in dose, the subjects are randomized to one of two treatment groups: either 2000 or 4000 IU/day to be taken throughout pregnancy until delivery.
  Interventions: Drug: cholecalciferol (vitamin D3); Drug: cholecalciferol
- Cholecalciferol 4000 IU (Experimental): Women are randomized to one of 2 treatment groups: 2000 or 4000 IU vitamin D3/day
  Interventions: Drug: cholecalciferol (vitamin D3); Drug: cholecalciferol

INTERVENTIONS:
Drug: cholecalciferol (vitamin D3) — randomized to one of two treatments: 2000 or 4000 IU vitamin D3/day
  Other Names: vitamin D3
Drug: cholecalciferol — randomized to one of 2 treatment doses: 2000 vs. 4000 IU/day vitamin D3
  Other Names: Vitamin D3
Drug: cholecalciferol — cholecalciferol at 2000 or 4000 IU/day to be taken througout pregnancy. This follows the initial run-in dosing of 2000 IU/day starting at 12-weeks' gestation.
  Other Names: Vitamin D3

SUMMARY:
Science News (October 2004) called vitamin D deficiency a "silent epidemic" in America, with no group unaffected. Using new guidelines of optimal vitamin D levels, more than 90% of African American women now suffer from vitamin D deficiency. Deficiency during pregnancy has profound effects on the developing fetus. Other systems besides bones are affected by vitamin D deficiency, including an increased risk of autoimmune diseases such as rheumatoid arthritis, multiple sclerosis, type I diabetes, and certain cancers.

This study proposes to examine and manage vitamin D levels in more than one thousand women in an underserved population in South Carolina. The women will be from the patient population seeking OB/GYN and Pediatric services through Eau Claire Cooperative Health Centers, Inc. (ECCHC), a network of ten clinics in three counties in the center of the state approximately 70 miles from Charleston, SC. ECCHC is one of approximately 1000 community health centers supported through Health and Human Services' (HHS) Health Resources and Services Administration's (HRSA), Bureau of Primary Health Care.

The research objectives for this project will be managed through the Pediatric Nutritional Sciences Research Center of the Children's Research Institute at the Medical University of South Carolina, Charleston, SC, in collaboration with ECCHC. The research aims will evaluate vitamin D levels and possible contributing factors to the levels in pregnant women. Women who present to ECCHC within the first trimester of pregnancy will be randomized to one of two doses of vitamin D supplementation shown to be effective in other groups. Each pregnant mother will begin supplementation during the 12th week of pregnancy and will be followed closely throughout pregnancy for one year to determine the effectiveness of supplementation on vitamin D status, overall health of mother, and of her infant following delivery.

We expect to observe severe vitamin D deficiency in a considerable percentage of the mothers and their infants who receive care at ECCHC, especially those individuals with darker pigmentation. When the extent of vitamin D deficiency within each racial/ethnic group is better defined and their supplementation requirements identified, we will be better able to establish guidelines for supplementation and health maintenance, and set policy recommendations for the dietary recommended intake of vitamin D. Those women and their infants identified as deficient in vitamin D will be important in establishing community health care policies for vitamin D surveillance and supplementation strategies. The results will allow us to implement specific dietary and/or medical interventions aimed at correcting hypovitaminosis D in the population in this study and other similar populations being served by the more than 1000 community health centers nationally.

DETAILED DESCRIPTION:
With avoidance of sunlight exposure due to lifestyle changes and concerns regarding skin cancer and the resultant widespread use of sunscreen, very few Americans are meeting their needs for vitamin D either through skin photosynthesis or dietary intake. A study published by the Centers for Disease Control (CDC) and our laboratory at the Medical University of South Carolina (MUSC) revealed that 42% of African American women in their childbearing years exhibited a deficiency of D vitamin (hypovitaminosis D) (1). Using new guidelines of optimal vitamin D levels, more than 90% of African American women now suffer from vitamin D deficiency (2). Science News (October 2004) called vitamin D deficiency a "silent epidemic" in America, with no group unaffected (3). Deficiency during pregnancy has profound effects on the developing fetus. Vitamin D deficiency affects other systems besides bones: it is associated with later, lifelong sequelae, with notable increased risk of autoimmune diseases such as rheumatoid arthritis (4), multiple sclerosis (5,6), type I diabetes (7,8), and certain cancers (7,9-14). Prevention and intervention studies only recently have been undertaken (3). A reexamination of dietary vitamin D requirements of various vulnerable populations in the U.S. is desperately needed (2,3). As a representative community with a diverse population, Eau Claire Cooperative Health Centers in South Carolina (ECCHC) serves a large percentage of African American as well as Caucasian and Hispanic women and children considered to be at high risk for vitamin D deficiency. ECCHC has eight clinics providing 1o care services to patients with special emphasis on Pediatric and OB/GYN services. Defining the prevalence of vitamin D deficiency in this patient population and the optimal vitamin D supplementation strategies for these women and their infants will become the prototype for recommendations applicable to other communities throughout the U.S.

In Specific Aim 1, the vitamin D status of a cross-sectional sample of 1000 pregnant women presenting at ECCHC for their prenatal care will be determined by measuring serum calcium, phosphorus, intact parathyroid hormone (iPTH), 25(OH)D, the nutritional marker of vitamin D as a function of ethnicity. Maternal health characteristics, skin pigmentation (using reflectance spectrophotometry), dietary characteristics (using an established food frequency questionnaire), and lifestyle profiles (using standardized questionnaires) will be ascertained as well. Any deficiency noted will lead to specific recommendations for vitamin D supplementation by the research team, with standardized strategies to monitor status following initiation of supplementation in Specific Aim 2. Based on extensive preliminary data, a supplementation regimen will be implemented and its efficacy in achieving optimal vitamin D status in these women tested in Aim 2: women within three racial groups (African American, Hispanic and Caucasian) will be stratified into two groups by their initial 25(OH)D level: Group 1, <32 ng/mL (less than optimal vitamin D status) and Group 2, ≥32 ng/mL (optimal vitamin D status). Based on our ongoing NIH study of pregnant women, each group will be randomized to receive one of two doses starting at 13 weeks' gestation: 2,000 or 4,000 IU vitamin D3/day after a universal one-month 2,000 IU/day dosing run-in period at 12 weeks' balanced by race/ethnicity. The randomization schema allows determination of both efficacy and safety for those deficient and those replete at entry into the study as a function of race/ethnicity and season.

Anticipated Results and Future Studies: We expect to observe vitamin D deficiency in a considerable percentage of the mothers and their newborn infants who receive care at ECCHC, especially those individuals with darker pigmentation. In Aims 1 & 2, by determining the prevalence of vitamin D deficiency with each racial/ethnic group, we will establish guidelines for supplementation and health maintenance, and policy recommendations for the dietary recommended intake of vitamin D in the U.S. The results will allow us to implement specific dietary and/or medical interventions aimed at correcting hypovitaminosis D in the population in this study and other similar populations being served by the more than 1000 community health centers nationally.

ELIGIBILITY:
Inclusion Criteria:

Aim 1: Any mother who presents to her obstetrician or midwife at Eau Claire with confirmation of a singleton pregnancy will be eligible for enrollment in Aim 1.

Aim 2: If the mother also is <12 completed weeks of gestation, she will be eligible for participation of Aim 2 of the study. Mothers of diverse ethnic background (African-American, Asian, Caucasian, Asian and Hispanic) actively will be recruited. There are no age exclusion criteria.

Exclusion Criteria:

Aim 1: There are no exclusion criteria.

Aim 2: Mothers with pre-existing calcium, parathyroid conditions or who require chronic diuretic or cardiac medication therapy including calcium channel blockers will not be eligible for enrollment into the study. Mothers with active thyroid disease (e.g., Graves, Hashimoto's or thyroiditis) will not be eligible to participate in the study; however, mothers on thyroid supplement with normal serological parameters may participate in the study if they are without any other endocrine dysfunction. Mothers with diabetes will not be excluded from participation in the study as vitamin D deficiency appears linked with insulin resistance and may aggravate the maternal condition.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 564 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Wagner, MD, Principal Investigator — Medical University of South Carolina; Stuart A Hamilton, M.D., Principal Investigator — Eau Claire Cooperative Health Centers
Locations (1):
- Eau Claire Cooperative Health Centers, Inc., Columbia, South Carolina, United States

REFERENCES:
- [Background] Hollis BW, Wagner CL. Vitamin D deficiency during pregnancy: an ongoing epidemic. Am J Clin Nutr. 2006 Aug;84(2):273. doi: 10.1093/ajcn/84.1.273. No abstract available. PMID 16895872
- [Background] Hollis BW, Wagner CL. Nutritional vitamin D status during pregnancy: reasons for concern. CMAJ. 2006 Apr 25;174(9):1287-90. doi: 10.1503/cmaj.060149. No abstract available. PMID 16636329
- [Background] Hollis BW, Wagner CL. Vitamin D requirements during lactation: high-dose maternal supplementation as therapy to prevent hypovitaminosis D for both the mother and the nursing infant. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1752S-8S. doi: 10.1093/ajcn/80.6.1752S. PMID 15585800
- [Result] Hamilton SA, McNeil R, Hollis BW, Davis DJ, Winkler J, Cook C, Warner G, Bivens B, McShane P, Wagner CL. Profound Vitamin D Deficiency in a Diverse Group of Women during Pregnancy Living in a Sun-Rich Environment at Latitude 32 degrees N. Int J Endocrinol. 2010;2010:917428. doi: 10.1155/2010/917428. Epub 2010 Dec 9. PMID 21197089
- See also: Thrasher Research Foundation — http://www.thrasherresearch.org/
- See also: Medical University of South Carolina, Charleston, SC — http://www.musc.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 564 women consented to participate in Aim 1 of the study (collection of cross-sectional baseline measures only). Of those 564 women, 265 were enrolled in Aim 2 of the study; only the Aim 2 cohort were randomized to intervention groups and followed through delivery.
Period: Overall Study
Arm/Group | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Started | 134 | 131
Completed | 72 | 66
Not Completed | 62 | 65

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU | Total
Number analyzed (Participants) | 134 | 131 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (5.5) | 25.2 (4.8) | 24.8 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 134 | 131 | 265
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 25-hydroxyvitamin D at Visit 7
Description: 25-hydroxyvitamin D at Visit 7, one month prior to delivery
Time Frame: 7 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Number analyzed (Participants) | 72 | 66
ng/mL | 36.7 (14.9) | 39.8 (12.9)

2. Secondary Outcome: Parathyroid Hormone at Visit 7
Description: Intact parathyroid hormone at Visit 7, one month prior to delivery
Time Frame: 7 months
Population: There was 1 subject in the 2000 IU group and 3 subjects in the 4000 IU group missing PTH measurements.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Number analyzed (Participants) | 71 | 63
pg/mL | 17.3 (8.3) | 14.3 (6.9)

ADVERSE EVENTS:
Arm/Group | Cholecalciferol 2000 IU | Cholecalciferol 4000 IU
Serious Adverse Events (participants affected / at risk) | 5/134 | 2/131
Other Adverse Events (participants affected / at risk) | 30/134 | 20/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol 2000 IU (N=134) | Cholecalciferol 4000 IU (N=131)
Fetal loss (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol 2000 IU (N=134) | Cholecalciferol 4000 IU (N=131)
Complications of Pregnancy (Pregnancy, puerperium and perinatal conditions) | 30 (30) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No